CLINICAL TRIAL: NCT02052232
Title: Study of Acute Muscle Protein Metabolism in Healthy Older Subjects
Brief Title: Study of Protein Metabolism in Healthy Older Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: BL19
Record Dates: First submitted 2013-12-06; First posted 2014-02-03 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Control protein powder sachet
  Interventions: Other: Control protein powder sachet
- Experimental (Experimental): Experimental protein powder sachet
  Interventions: Other: Experimental protein powder sachet

INTERVENTIONS:
Other: Experimental protein powder sachet — mixed with 8 oz. water
  Arms: Experimental
Other: Control protein powder sachet — mixed with 8 oz. water
  Arms: Control

SUMMARY:
This is a randomized, double-blinded, crossover study to evaluate muscle protein metabolism during fasting and feeding in healthy older subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 and ≤ 75 years
* Body Mass Index (BMI) > 23.0 to < 30.0
* Ability (with or without the aid of an assistive device) to climb a flight of 10 stairs or walk an equivalent of 1 city block without assistance
* Currently not participating in a formal exercise or training program and agrees to refrain from intense physical activity from screening through the completion of the study.

Exclusion Criteria:

* Diagnosis of diabetes
* Active pursuit of weight loss
* Poorly controlled hypertension or hypotension
* Untreated hypothyroidism or hyperthyroidism
* Anemia or abnormally functioning kidneys or liver
* A significant cardiovascular event within ≤ 6 months; or stated history of congestive heart failure; or evidence of clinically active cardiovascular disease assessed during the screening EKG
* Peripheral arterial disease or other diseases that preclude proper limb blood flow
* Chronic, contagious, infectious disease
* Current infection or corticosteroid treatment within the last 3 months
* Clotting or bleeding disorders, stated history of Deep Vein Thrombosis (DVT) and/or a known hypercoagulable condition
* In condition deemed unsuitable for study based upon study physician assessment
* Surgery requiring >2 days of hospitalization in the last 3 weeks and/or planned elective surgery requiring >2 days of hospitalization during the course of the study
* Current active malignant disease or was treated within the last 6 months for cancer
* An amputee
* Obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease
* Diagnosed with, or has a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse
* Cannot refrain from taking

  * High doses of fish oil, or omega-3 supplements, or high doses of vitamin D
  * Medications/dietary supplements/herbals or substances that are considered anabolic, or reduce weight
  * Any pulmonary anti-inflammatory medication or bronchodilators on the day of and 48 hours prior to study visits 1 and 2
  * NSAIDS or acetaminophen on the day of and 48 hours prior to study visits 1 and 2
* Chronic use of nicotine
* Allergic or intolerant to any ingredient found in the study products

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Protein Metabolism | Change from - 1 to + 5 hours
  Study Visit 1 and Study Visit 2

SECONDARY OUTCOMES:
Macrovascular Blood Flow | Change from -1 to +5 hours
  Study Visit 1 and Study Visit 2
Glycemic Markers | Change from -1 to +5 hours
  Study Visit 1 and Study Visit 2
Microvascular Blood Flow | Change from -1 to +5 hours
  Study Visit 1 and Study Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Min Tian, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Nottingham, Derby, United Kingdom